CLINICAL TRIAL: NCT01848496
Title: A Double-blind Randomized Clinical Trial of Two Techniques for Gingival Displacement
Brief Title: Clinical Trial of Two Techniques for Gingival Displacement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maximiliano Sergio Cenci (Other)
Responsible Party: Sponsor-Investigator, Maximiliano Sergio Cenci, Professor, Federal University of Pelotas
Organization: Federal University of Pelotas (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO0015
Record Dates: First submitted 2013-04-25; First posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Poor Aesthetic of Existing Restoration of Tooth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cordless technique (Experimental): This technique does not employ a gingival cord to obtain gingival displacement.
  Interventions: Procedure: Gingival displacement
- Conventional technique (Active Comparator): This technique employ a gingival cord to obtain gingival displacement.
  Interventions: Procedure: Gingival displacement

INTERVENTIONS:
Procedure: Gingival displacement — Gingival displacement is a dental procedure that allows exposure of the finishing line of a dental cavity in order to produce a well-adapted restoration.

SUMMARY:
Regardless of the selected technique for dental impression, gingival displacement is an essential procedure specially when making impressions of subgingival finishing lines, because a moisture-free sulcus is a requirement for an effective impression.

The objective of this randomized clinical study is to evaluate the efficacy of the conventional and cordless gingival displacement (GD) techniques.

DETAILED DESCRIPTION:
On conventional technique we normally use a cord for gingival displacement. On the other hand, on cordless technique do not require this need.

ELIGIBILITY:
Inclusion Criteria:

* good general and dental health
* at least two anterior teeth with an indication of prosthetic dental crown

Exclusion Criteria:

* smoking habits
* systemic diseases
* pregnant
* had not consumed antibiotics or anti-inflammatory drugs in the last 60 days
* the selected teeth must have good periodontal health characterized by regular gingival margin with at least 2 mm of attached gingiva, non-fibrotic gingival tissue, no marginal recession, probing depth ≤ 3 mm, no evidence of significant loss of bone insertion and present no visible plaque and gingival bleeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Interleukins concentration on gingival crevicular fluid | Before and 1 day after gilgival displacement

SECONDARY OUTCOMES:
Periodontal indices | Before, 1 day after and 10 day after gingival displacement
  Periodontal indices (attachment level, gingival bleeding and plaque index) were evaluated before and after gingival displacement by the both techniques.

OTHER OUTCOMES:
Self-reported unpleasant flavour and pain | Immediatelly after interventions
  Also were evaluated subjective parameters (unpleasant flavor and pain) self-reported by the volunteers during gingival displacement. These subjective outcomes were collected using the visual analogic scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo R Sarmento, MSc, Study Chair — Federal University of Pelotas; Fernanda Faot, PhD, Principal Investigator — Federal University of Pelotas; Fábio RM Leite, PhD, Study Director — Federal University of Pelotas
Locations (1):
- Pelotas Dental School, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Al Hamad KQ, Azar WZ, Alwaeli HA, Said KN. A clinical study on the effects of cordless and conventional retraction techniques on the gingival and periodontal health. J Clin Periodontol. 2008 Dec;35(12):1053-8. doi: 10.1111/j.1600-051X.2008.01335.x. PMID 19040582
- [Background] Passariello C, Puttini M, Virga A, Gigola P. Microbiological and host factors are involved in promoting the periodontal failure of metaloceramic crowns. Clin Oral Investig. 2012 Jun;16(3):987-95. doi: 10.1007/s00784-011-0585-0. Epub 2011 Jul 1. PMID 21720749
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834